CLINICAL TRIAL: NCT00978055
Title: Single-Dose Fasting Bioequivalence Study of Liothyronine Sodium Tablets (50 Mcg; Mylan) to Cytomel® Tablets (50 Mcg; King) in Healthy Euthyroid Adult Volunteers
Brief Title: Fasting Study of Liothyronine Sodium Tablets (50 Mcg) to Cytomel® Tablets (50 Mcg)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Wayne Talton, Mylan, Inc.
Organization: MylanPharma (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: LIOT-0592
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Healthy

ARMS (2):
- 1 (Experimental): Liothyronine Sodium Tablets, 50 mcg
  Interventions: Drug: 1: Liothyronine Sodium Tablets
- 2 (Active Comparator): Cytomel® Tablets, 50 mcg
  Interventions: Drug: 2: Cytomel® Tablets

INTERVENTIONS:
Drug: 1: Liothyronine Sodium Tablets — Liothyronine Sodium Tablets, 50 mcg
  2 x 50 mcg, single-dose, fasting
  Arms: 1
Drug: 2: Cytomel® Tablets — Cytomel® Tablets, 50 mcg
  2 x 50 mcg, single-dose, fasting
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's liothyronine sodium 50 mcg tablets to King's Cytomel® 50 mcg tablets following a single, oral 100 mcg (2 x 50 mcg) dose administration under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy males and/or non-pregnant, non-lactating females, 18 years and older
* able to swallow medication

Exclusion Criteria:

* institutionalized subjects
* history of any significant disease
* use of any prescription or OTC medications within 14 days prior to start of study
* received any investigational products within 30 days prior to start of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com